CLINICAL TRIAL: NCT03925597
Title: Multiomic Signatures of Microbial Metabolites Following Prebiotic Fiber Supplementation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael Snyder, Chairman and Professor of Genetics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 23602; 5R01AT010232 (NIH)
Record Dates: First submitted 2018-12-20; First posted 2019-04-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-04

CONDITIONS: Prebiotics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the order of the fiber supplementation and they will take each fiber for three weeks. After a washout period, they will switch fibers. Blood and stool samples will be collected through the intervention and once during each washout period.
Who Masked: Participant
Masking Description: Participant will be given the unlabeled fiber supplement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (24):
- ARM 1: Arabinoxylan, Beta-Glucan, Resistant Starch, Inulin (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Arabinoxylan, Beta-Glucan, Resistant Starch, Inulin.
  Interventions: Dietary Supplement: Fiber cycles ARM 1
- ARM 2: Arabinoxylan, Beta-Glucan, Inulin, Resistant Starch (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Arabinoxylan, Beta-Glucan, Inulin, Resistant Starch.
  Interventions: Dietary Supplement: Fiber cycles ARM 2
- ARM 3: Arabinoxylan, Resistant Starch, Beta-Glucan, Inulin (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: rabinoxylan, Resistant Starch, Beta-Glucan, Inulin.
  Interventions: Dietary Supplement: Fiber cycles ARM 3
- ARM 4: Arabinoxylan, Resistant Starch, Inulin, Beta-Glucan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Arabinoxylan, Resistant Starch, Inulin, Beta-Glucan.
  Interventions: Dietary Supplement: Fiber cycles ARM 4
- ARM 5: Arabinoxylan, Inulin, Beta-Glucan, Resistant Starch (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Arabinoxylan, Inulin, Beta-Glucan, Resistant Starch.
  Interventions: Dietary Supplement: Fiber cycles ARM 5
- ARM 6: Arabinoxylan, Inulin, Resistant Starch, Beta-Glucan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Arabinoxylan, Inulin, Resistant Starch, Beta-Glucan.
  Interventions: Dietary Supplement: Fiber cycles ARM 6
- ARM 7: Beta-Glucan, Arabinoxylan, Resistant Starch, Inulin (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Beta-Glucan, Arabinoxylan, Resistant Starch, Inulin.
  Interventions: Dietary Supplement: Fiber cycles ARM 7
- ARM 8: Beta-Glucan, Arabinoxylan, Inulin, Resistant Starch (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Beta-Glucan, Arabinoxylan, Inulin, Resistant Starch.
  Interventions: Dietary Supplement: Fiber cycles ARM 8
- ARM 9: Beta-Glucan, Resistant Starch, Inulin, Arabinoxylan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Beta-Glucan, Resistant Starch, Inulin, Arabinoxylan.
  Interventions: Dietary Supplement: Fiber cycles ARM 9
- ARM 10: Beta-Glucan, Resistant Starch, Arabinoxylan, Inulin (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Beta-Glucan, Resistant Starch, Arabinoxylan, Inulin.
  Interventions: Dietary Supplement: Fiber cycles ARM 10
- ARM 11: Beta-Glucan, Inulin, Arabinoxylan, Resistant Starch (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Beta-Glucan, Inulin, Arabinoxylan, Resistant Starch.
  Interventions: Dietary Supplement: Fiber cycles ARM 11
- ARM 12: Beta-Glucan, Inulin, Resistant Starch, Arabinoxylan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Beta-Glucan, Inulin, Resistant Starch, Arabinoxylan.
  Interventions: Dietary Supplement: Fiber cycles ARM 12
- ARM 13: Resistant Starch, Inulin, Beta-Glucan, Arabinoxylan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Resistant Starch, Inulin, Beta-Glucan, Arabinoxylan.
  Interventions: Dietary Supplement: Fiber cycles ARM 13
- ARM 14: Resistant Starch, Inulin, Arabinoxylan, Beta-Glucan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Resistant Starch, Inulin, Arabinoxylan, Beta-Glucan.
  Interventions: Dietary Supplement: Fiber cycles ARM 14
- ARM 15: Resistant Starch, Arabinoxylan, Inulin, Beta-Glucan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Resistant Starch, Arabinoxylan, Inulin, Beta-Glucan.
  Interventions: Dietary Supplement: Fiber cycles ARM 15
- ARM 16: Resistant Starch, Arabinoxylan, Beta-Glucan, Inulin (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Resistant Starch, Arabinoxylan, Beta-Glucan, Inulin.
  Interventions: Dietary Supplement: Fiber cycles ARM 16
- ARM 17: Resistant Starch, Beta-Glucan, Inulin, Arabinoxylan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Resistant Starch, Beta-Glucan, Inulin, Arabinoxylan.
  Interventions: Dietary Supplement: Fiber cycles ARM 17
- ARM 18: Resistant Starch, Beta-Glucan, Arabinoxylan, Inulin (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Resistant Starch, Beta-Glucan, Arabinoxylan, Inulin.
  Interventions: Dietary Supplement: Fiber cycles ARM 18
- ARM 19: Inulin, Resistant Starch, Arabinoxylan, Beta-Glucan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Inulin, Resistant Starch, Arabinoxylan, Beta-Glucan.
  Interventions: Dietary Supplement: Fiber cycles ARM 19
- ARM 20: Inulin, Resistant Starch, Beta-Glucan, Arabinoxylan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Inulin, Resistant Starch, Beta-Glucan, Arabinoxylan.
  Interventions: Dietary Supplement: Fiber cycles ARM 20
- ARM 21: Inulin, Beta-Glucan, Resistant Starch, Arabinoxylan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Inulin, Beta-Glucan, Resistant Starch, Arabinoxylan.
  Interventions: Dietary Supplement: Fiber cycles ARM 21
- ARM 22: Inulin, Beta-Glucan, Arabinoxylan, Resistant Starch (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Inulin, Beta-Glucan, Arabinoxylan, Resistant Starch.
  Interventions: Dietary Supplement: Fiber cycles ARM 22
- ARM 23: Inulin, Arabinoxylan, Beta-Glucan, Resistant Starch (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Inulin, Arabinoxylan, Beta-Glucan, Resistant Starch.
  Interventions: Dietary Supplement: Fiber cycles ARM 23
- ARM 24: Inulin, Arabinoxylan, Resistant Starch, Beta-Glucan (Experimental): Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks. In this arm, participants will take the fiber supplements in the following order: Inulin, Arabinoxylan, Resistant Starch, Beta-Glucan.
  Interventions: Dietary Supplement: Fiber cycles ARM 24

INTERVENTIONS:
Dietary Supplement: Fiber cycles ARM 1 — Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Arabinoxylan. On cycle 2, they will take 20g per day of Beta-Glucan. On cycle 3, they will take 20g per day of Resistant Starch. On cycle 4, they will take 20g per day of Inulin.
  Arms: ARM 1: Arabinoxylan, Beta-Glucan, Resistant Starch, Inulin
Dietary Supplement: Fiber cycles ARM 2 — Participants will complete 4 cycles. For each cycle they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Arabinoxylan. On cycle 2, they will take 20g per day of Beta-Glucan. On cycle 3, they will take 20g per day of Inulin. On cycle 4, they will take 20g per day of Resistant Starch.
  Arms: ARM 2: Arabinoxylan, Beta-Glucan, Inulin, Resistant Starch
Dietary Supplement: Fiber cycles ARM 3 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Arabinoxylan. On cycle 2, they will take 20g per day of Resistant Starch. On cycle 3, they will take 20g per day of Beta-Glucan. On cycle 4, they will take 20g per day of Inulin.
  Arms: ARM 3: Arabinoxylan, Resistant Starch, Beta-Glucan, Inulin
Dietary Supplement: Fiber cycles ARM 4 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Arabinoxylan. On cycle 2, they will take 20g per day of Resistant Starch. On cycle 3, they will take 20g per day of Inulin. On cycle 4, they will take 20g per day of Beta-Glucan.
  Arms: ARM 4: Arabinoxylan, Resistant Starch, Inulin, Beta-Glucan
Dietary Supplement: Fiber cycles ARM 5 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Arabinoxylan. On cycle 2, they will take 20g per day of Inulin. On cycle 3, they will take 20g per day of Beta-Glucan. On cycle 4, they will take 20g per day of Resistant Starch.
  Arms: ARM 5: Arabinoxylan, Inulin, Beta-Glucan, Resistant Starch
Dietary Supplement: Fiber cycles ARM 6 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Arabinoxylan. On cycle 2, they will take 20g per day of Inulin. On cycle 3, they will take 20g per day of Resistant Starch. On cycle 4, they will take 20g per day of Beta-Glucan.
  Arms: ARM 6: Arabinoxylan, Inulin, Resistant Starch, Beta-Glucan
Dietary Supplement: Fiber cycles ARM 7 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Beta-Glucan. On cycle 2, they will take 20g per day of Arabinoxylan. On cycle 3, they will take 20g per day of Resistant Starch. On cycle 4, they will take 20g per day of Inulin.
  Arms: ARM 7: Beta-Glucan, Arabinoxylan, Resistant Starch, Inulin
Dietary Supplement: Fiber cycles ARM 8 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Beta-Glucan. On cycle 2, they will take 20g per day of Arabinoxylan. On cycle 3, they will take 20g per day of Inulin. On cycle 4, they will take 20g per day of Resistant Starch.
  Arms: ARM 8: Beta-Glucan, Arabinoxylan, Inulin, Resistant Starch
Dietary Supplement: Fiber cycles ARM 9 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Beta-Glucan. On cycle 2, they will take 20g per day of Resistant Starch. On cycle 3, they will take 20g per day of Inulin. On cycle 4, they will take 20g per day of Arabinoxylan.
  Arms: ARM 9: Beta-Glucan, Resistant Starch, Inulin, Arabinoxylan
Dietary Supplement: Fiber cycles ARM 10 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Beta-Glucan. On cycle 2, they will take 20g per day of Resistant Starch. On cycle 3, they will take 20g per day of Arabinoxylan. On cycle 4, they will take 20g per day of Inulin.
  Arms: ARM 10: Beta-Glucan, Resistant Starch, Arabinoxylan, Inulin
Dietary Supplement: Fiber cycles ARM 11 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Beta-Glucan. On cycle 2, they will take 20g per day of Inulin. On cycle 3, they will take 20g per day of Arabinoxylan. On cycle 4, they will take 20g per day of Resistant Starch.
  Arms: ARM 11: Beta-Glucan, Inulin, Arabinoxylan, Resistant Starch
Dietary Supplement: Fiber cycles ARM 12 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Beta-Glucan. On cycle 2, they will take 20g per day of Inulin. On cycle 3, they will take 20g per day of Resistant Starch. On cycle 4, they will take 20g per day of Arabinoxylan.
  Arms: ARM 12: Beta-Glucan, Inulin, Resistant Starch, Arabinoxylan
Dietary Supplement: Fiber cycles ARM 13 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Resistant Starch. On cycle 2, they will take 20g per day of Inulin. On cycle 3, they will take 20g per day of Beta-Glucan. On cycle 4, they will take 20g per day of Arabinoxylan.
  Arms: ARM 13: Resistant Starch, Inulin, Beta-Glucan, Arabinoxylan
Dietary Supplement: Fiber cycles ARM 14 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Resistant Starch. On cycle 2, they will take 20g per day of Inulin. On cycle 3, they will take 20g per day of Arabinoxylan. On cycle 4, they will take 20g per day of Beta-Glucan.
  Arms: ARM 14: Resistant Starch, Inulin, Arabinoxylan, Beta-Glucan
Dietary Supplement: Fiber cycles ARM 15 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Resistant Starch. On cycle 2, they will take 20g per day of Arabinoxylan. On cycle 3, they will take 20g per day of Inulin. On cycle 4, they will take 20g per day of Beta-Glucan.
  Arms: ARM 15: Resistant Starch, Arabinoxylan, Inulin, Beta-Glucan
Dietary Supplement: Fiber cycles ARM 16 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Resistant Starch. On cycle 2, they will take 20g per day of Arabinoxylan. On cycle 3, they will take 20g per day of Beta-Glucan. On cycle 4, they will take 20g per day of Inulin.
  Arms: ARM 16: Resistant Starch, Arabinoxylan, Beta-Glucan, Inulin
Dietary Supplement: Fiber cycles ARM 17 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Resistant Starch. On cycle 2, they will take 20g per day of Beta-Glucan. On cycle 3, they will take 20g per day of Inulin. On cycle 4, they will take 20g per day of Arabinoxylan.
  Arms: ARM 17: Resistant Starch, Beta-Glucan, Inulin, Arabinoxylan
Dietary Supplement: Fiber cycles ARM 18 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Resistant Starch. On cycle 2, they will take 20g per day of Beta-Glucan. On cycle 3, they will take 20g per day of Arabinoxylan. On cycle 4, they will take 20g per day of Inulin.
  Arms: ARM 18: Resistant Starch, Beta-Glucan, Arabinoxylan, Inulin
Dietary Supplement: Fiber cycles ARM 19 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Inulin. On cycle 2, they will take 20g per day of Resistant Starch. On cycle 3, they will take 20g per day of Arabinoxylan. On cycle 4, they will take 20g per day of Beta-Glucan.
  Arms: ARM 19: Inulin, Resistant Starch, Arabinoxylan, Beta-Glucan
Dietary Supplement: Fiber cycles ARM 20 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Inulin. On cycle 2, they will take 20g per day of Resistant Starch. On cycle 3, they will take 20g per day of Beta-Glucan. On cycle 4, they will take 20g per day of Arabinoxylan.
  Arms: ARM 20: Inulin, Resistant Starch, Beta-Glucan, Arabinoxylan
Dietary Supplement: Fiber cycles ARM 21 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Inulin. On cycle 2, they will take 20g per day of Beta-Glucan. On cycle 3, they will take 20g per day of Resistant Starch. On cycle 4, they will take 20g per day of Arabinoxylan.
  Arms: ARM 21: Inulin, Beta-Glucan, Resistant Starch, Arabinoxylan
Dietary Supplement: Fiber cycles ARM 22 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Inulin. On cycle 2, they will take 20g per day of Beta-Glucan. On cycle 3, they will take 20g per day of Arabinoxylan. On cycle 4, they will take 20g per day of Resistant Starch.
  Arms: ARM 22: Inulin, Beta-Glucan, Arabinoxylan, Resistant Starch
Dietary Supplement: Fiber cycles ARM 23 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Inulin. On cycle 2, they will take 20g per day of Arabinoxylan. On cycle 3, they will take 20g per day of Beta-Glucan. On cycle 4, they will take 20g per day of Resistant Starch.
  Arms: ARM 23: Inulin, Arabinoxylan, Beta-Glucan, Resistant Starch
Dietary Supplement: Fiber cycles ARM 24 — Participants will complete 4 cycles. For each cycle, they will take 20g per day fiber supplement for 3 weeks, followed by a washout period of at least 6-8 weeks.
  On cycle 1, they will take 20g per day of Inulin. On cycle 2, they will take 20g per day of Arabinoxylan. On cycle 3, they will take 20g per day of Resistant Starch. On cycle 4, they will take 20g per day of Beta-Glucan.
  Arms: ARM 24: Inulin, Arabinoxylan, Resistant Starch, Beta-Glucan

SUMMARY:
The investigators propose a comprehensive, multiomic study that will integrate longitudinal data associating changes in specific gut bacteria and host in response to prebiotic fiber supplementation. These data will guide the development of an integrative biological signature relating bacterial-derived metabolites with biological outcome in the host. The open sharing of data generated by the proposed research represents a significant public resource that will support and accelerate future novel studies.

DETAILED DESCRIPTION:
Phenolics-rich prebiotic fiber has been correlated with a number of positive health outcomes, however their bioavailability is typically low. A large portion the gut microbiota metabolize these fibers releasing a range of phenolic acids, which are believed to be principle bioactive components driving reduction in disease risk. Despite this, little evidence exists linking specific gut bacteria with the metabolites they produce and the downstream biological effects that these compounds exert. With this study, the investigators propose to assemble a cohort of healthy individuals that will receive prebiotic supplementation, during comprehensive, longitudinal characterization of the microbiota and host changes with clinical markers and multiple omics assays. These multiomic data will then be integrated, generating unique biological signatures that define the role that microbial metabolites from specific bacteria play in host biological activity. To validate the biological function of these microbial metabolites, gnobiotic mice will be inoculated with the microbial strains identified. The newly identified metabolites will also be synthesized in vitro to demonstrate their structure, biological properties and applications. Through this study the investigators expect to gain a detailed and clear understanding of the physiological changes, at the mechanistic level, that occur in the microbiome and host in response to dietary supplementation with prebiotic fiber.

ELIGIBILITY:
Inclusion Criteria:

- good general health

Exclusion Criteria:

* Chronic inflammatory conditions
* Major organ disease
* Heavy alcohol use
* Pregnancy/lactation
* Use of medication known to affect carbohydrate or lipid metabolism
* Active eating disorder

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Mapping of microbiota changes in response to prebiotic intervention | 3 years
  A detailed map of microbes and microbial gene expression changes during the intervention will be developed.
  Microbiota complexity in fecal samples will be determined by shotgun metagenomic sequencing. Novel microbes and gene pathways will be identified by de novo assemble of whole fecal metagenomes.
Comprehensive phenotyping of host profile during prebiotic intervention | 4 years
  Changes in host (human) phenotypic profile during the prebiotic intervention will be determined.
  Profile will include the metagenome, transcriptome, metabolome and cytokines of participants during the prebiotic intervention.
Biological signatures identified from the integration of microbiome-host omes | 4 years
  Biological signatures will be developed from the integration of the omics data with microbial metabolite levels.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Snyder, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No